CLINICAL TRIAL: NCT00384696
Title: Health Communications and Risk Processing Among Smokers
Brief Title: Risk Perception Among Quitting Smokers
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2004-0806; 1 K01 CD000193-01 (Other: NCI)
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Smoking
Keywords: Risk Perception; Smoking Cessation; Nicotine Replacement Therapy; Questionnaire; Nicotine
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Nicotine Replacement Therapy; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Smoking Cessation: Treatment to help quit smoking, including written self-help materials, counseling, and 4 week supply of nicotine patch plus 5 MD Anderson Visits.
  Interventions: Drug: Nicotine Replacement Therapy; Behavioral: Questionnaire

INTERVENTIONS:
Drug: Nicotine Replacement Therapy — 4 Weeks of nicotine patch. Patch therapy for participants who smoke >10 cigarettes/day consists of 2 weeks of 21 mg patches, 1 week of 14 mg patches, and 1 week of 7 mg patches. Patch therapy for participants who smoke 5-10 cigarettes/day consists of 2 weeks of 14 mg patches and 2 weeks of 7 mg patches.
Behavioral: Questionnaire — Survey taking 1 and 1/2 hours at each study visit.

SUMMARY:
The goal of this behavioral research study is to put together and study a treatment for nicotine dependence that looks at how participant's thoughts and feelings about smoking may be related to how successfully they quit smoking.

DETAILED DESCRIPTION:
If patient agrees to participate, they will receive free treatment to help them quit smoking, including written self-help materials, counseling, and a supply of the nicotine patch for 4 weeks. Participant will visit M. D. Anderson 5 times during this study; once for an orientation/intake visit, and then for 4 more study visits.

At the first (orientation) visit, participant will be asked about their feelings and moods, as well as their smoking status. Participant will fill out questionnaires on a computer and complete a breath test. The questionnaires will be about mood, stress, and smoking-related issues, and should take about 1 hour and 30 minutes to complete. To complete the breath test, participant will blow into a tube that's attached to a machine about the size of a pocket computer. The breath test is used to estimate the amount of tobacco smoke that participant inhales. Participant will also complete two computer-based tasks. Women who are pregnant should not take part in this study.

In addition, participant will receive a palmtop personal computer and be trained in how to use it. Participant will carry this small computer with them from the time of their first visit until their last study visit. Participant will use the computer to answer questions about their mood, stress, and smoking-related issues. Participant will be asked to fill out some questions on the computer each time they have an urge to smoke or they actually smoke. Also, the computer will "beep" at random and set times and request that participant answers some questions.

Participant will return for 4 visits after the orientation session. During these visits, participant will receive brief individual counseling where they will discuss techniques to help them quit smoking. Participant will also be asked to fill out questionnaires on a computer about their moods and feelings, as well as their smoking status. The questionnaires should take about 30 minutes to complete. The breath test will be given at every clinic visit.

Participant may be contacted by mail, telephone, and/or e-mail throughout the study and follow-up period, to provide reminders of clinic visits. Participant may also be asked for information about their smoking status during the usual reminder calls and/or calls to reschedule missed appointments.

A supply of the nicotine patch will be provided to participant at each counseling session. The final supply of the patch is provided at the final counseling session.

This is an investigational study. The nicotine patch used in this study is approved by the Food and Drug Administration (FDA). About 20 people will take part in a pilot phase of this study; then, another 200 participants will take part in the main study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years.
2. Current smoker with a history of at least 5 cigarettes/day for the last year
3. Motivated to quit within the next week.
4. Home address and a functioning home telephone number.
5. Can speak, read, and write in English at a sixth-grade literacy level.

Exclusion Criteria:

1. Contraindication for nicotine patch use.
2. Active substance abuse or dependence.
3. Regular use of tobacco products other than cigarettes (cigars, pipes, smokeless).
4. Use of bupropion or nicotine products other than the nicotine patches supplied by the study.
5. Pregnancy or lactation.
6. Another household member enrolled in the study.
7. Participation in a smoking cessation program or study during the past 90 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Current smoker, age 18 to 65 years, with history of 5 cigarettes/day for last year wishing to quit
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2006-02-10 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk Perceptions Over Time Among Smokers and Non Smokers | 4 weeks
  Primary hypothesis is that abstainers will show higher risk perceptions than relapsers.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna H. McNeill, PHD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org